CLINICAL TRIAL: NCT05917639
Title: CommunICation of bEnefit Risk Information: an Online Randomised Controlled Trial
Acronym: CICERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R86270/RE001
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Knowledge, Attitudes, Practice; Literacy; Confidence, Self
Keywords: shared decision-making
MeSH Terms: conditions — Behavior; Literacy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitruvian plot (Experimental)
  Interventions: Device: Vitruvian plot
- Kilim plot (Experimental)
  Interventions: Device: Kilim plot
- Summary of findings table (Active Comparator)
  Interventions: Device: Summary of findings table

INTERVENTIONS:
Device: Vitruvian plot — Visual (magnitude, uncertainty) and written (magnitude) communication tool / interventional decision-making aid tool
  Arms: Vitruvian plot
Device: Kilim plot — Visual (uncertainty) and written (magnitude) communication tool / interventional decision-making aid tool
  Arms: Kilim plot
Device: Summary of findings table — Written (magnitude, uncertainty) communication tool / interventional decision-making aid tool
  Arms: Summary of findings table

SUMMARY:
How health-related information is communicated affects what is understood and might influence how people make decisions and how confident they feel in participating in clinical shared decision-making.

The CICERO trial will compare three different communication tools providing information on fictional interventions for a common medical problem (i.e. social anxiety disorder) both in terms of how well interventions work (benefit) and also possible harms associated (risk). The three communication tools ("Summary of Findings table", "Kilim plot", and "Vitruvian plot") differ in how they present information: exclusively written, primarily written and partially graphical, or mixed written and visual. Each participant will be asked to go through one clinical scenario.

The investigators will ask participants to familiarise themselves with the tool they have been allocated to (either a plot or a table) and then answer some validated questionnaires to measure how useful and efficient the communication strategy was.

The entire study occurs online in a single study session (about 20 minutes).

The results of the CICERO trial will inform how to communicate research findings to the general population, facilitating their implementation in clinical shared decision-making.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years (inclusive)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2178 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale, low literacy version | through study completion, an average of 20 minutes
  Higher scores indicate worse outcomes (min = 0; max = 100).

SECONDARY OUTCOMES:
Decision Self-Efficacy scale | through study completion, an average of 20 minutes
  Higher scores indicate better outcomes (min = 0; max = 100).
Preparation for Decision Making scale | through study completion, an average of 20 minutes
  Higher scores indicate better outcomes (min = 0; max = 100).
Information comprehension (proportion of participants providing a correct answer) | through study completion, an average of 20 minutes
  Participants will be asked to choose one of multiple (fictional) medical interventions based on their characteristics as part of the clinical scenario. The question related to the clinical scenario allows only one correct answer.

OTHER OUTCOMES:
Number of minutes to complete the questionnaire | through study completion, an average of 20 minutes
  Automated measurement from the first access to the online questionnaire (first input) to its completion (last input), assessed up to the end of the study (continuous outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Precision Psychiatry Lab (OxPPL), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CICERO trial — https://www.psych.ox.ac.uk/research/evidence-based-mental-health/cicero